CLINICAL TRIAL: NCT05031962
Title: Porcine Acellular Dermal Matrix (PADM)-Assisted Implant-based Breast Reconstruction: a Prospective Observational Study
Brief Title: Safety and Clinical Performance of a Biological Matrix Used in Implant-based Breast Reconstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Meccellis Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: BR_01_CIP
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Breast Reconstruction Following Mastectomy
Keywords: Breast reconstruction; Biological membrane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CELLIS Breast (Porcine Acellular Dermal Matrix, PADM): Implant-based breast reconstruction following mastectomy using the CELLIS Breast matrix
  Interventions: Device: CELLIS Breast (Porcine Acellular Dermal Matrix, PADM)

INTERVENTIONS:
Device: CELLIS Breast (Porcine Acellular Dermal Matrix, PADM) — Biological membrane used in breast reconstruction

SUMMARY:
The general objective of the study is to confirm the medium/long-term safety and clinical performance of the CELLIS Breast membranes used in breast reconstruction and to identify emerging risks in comparison to clinical data related to other treatment modalities.

The present study will be a prospective, multicentric, non-randomized and non-controlled trial involving 112 patients followed for 24 months. The study will be conducted in France in 7 investigational centres.

DETAILED DESCRIPTION:
The study will be prospective, multicentric, single-arm observational (non-interventional) to evaluate the safety and performance of the CELLIS Breast membranes used in breast reconstruction following mastectomy.

All evaluations will be performed and products used according to the usual practice, without additional or unusual diagnostic, treatment and monitoring procedure.

The study will be conducted in France in 7 investigational centres including 112 patients scheduled for a breast reconstruction following mastectomy.

Each patient will participate in one assessment period including a preoperative visit, followed by the day of surgical procedure and a hospitalization period.

Patients will return for ambulatory visits on day 10 (+/- 5 days) and/or on day 30 (+/- 7 days), on month 3 (+/- 2 weeks), on month 12 (+/- 2 weeks) and on month 24 (+/-2 weeks) post-surgery.

CELLIS Breast is available in one thickness, in a variety of size and forms addressing multiple surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥18 years,
* Patient with an indication of breast reconstruction after mastectomy (therapeutic or prophylactic),
* Patient being informed of her participation to the study and of the follow-up visits, and having no objection to the clinical data collection and medical file access,
* Patient being informed of the porcine origin of the device in advance of the procedure.

Exclusion Criteria:

* Patient with known hypersensitivity to porcine materials,
* Patient with an existing infection at the site of implantation,
* Patient having refused to participate to the study,
* Patient refusing to return for the follow-up visits,
* Patient who is pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Constitution and follow-up of a consecutive cohort of patients operated with the CELLIS Breast membranes based on the usual practices, the indication and the inclusion-exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events. Main complications of interest: infection, cellulitis, seroma, hematoma, skin flap-nipple necrosis, delayed wound healing, wound dehiscence, red breast syndrome, capsular contracture, implant related | From the surgical procedure throughout the entire 24-month follow-up period
  Percentage

SECONDARY OUTCOMES:
Patient aesthetic evaluation evaluated by Visual Analog Scale (VAS). The suppleness of the reconstruction will be evaluated (natural-hard): VAS score from 1 to 10 (1=very bad suppleness, breast hard; 10=excellent suppleness-natural breast). | At the 3, 12 and 24-month follow-up visits
  Described at each visit
Surgeon aesthetic evaluation: satisfaction related to the quality of the reconstruction (very good, good, fair, bad), suppleness (Visual Analog Scale score from 1 to 10 with 10=excellent suppleness) and symmetry (very good, good, fair, bad). | At the 3, 12 and 24-month follow-up visits
  Percentage of each modality and VAS score described at each visit
Patient-reported pain using a visual analogue scale (VAS) scored from 0 to 10 (0=no pain; 10=worse pain). | At the 10-day, 30-day, 3-month, 12-month and 24-month follow-up visits
  Described at each visit
Patient analgesics consumption | At the 10-day, 30-day, 3-month, 12-month and 24-month follow-up visits
  Percentage of analgesics consumption with a Cochrane-Armitage trend test.
Quality of life (QoL) by the use of the SF-36 questionnaire. | At baseline and at 24 month
  Change from screening of each domain score and total score at 24-month. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 with lower scores = more disability, and higher scores = less disability
Description of device deficiency: inadequacy of a medical device with respects to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequate labelling. | During the surgical procedure
  Summarized and listed

CONTACTS AND LOCATIONS:
Overall Officials: Michael ATLAN, MD, Principal Investigator — Hôpital Tenon, Paris, France
Locations (10):
- France (10):
  - Institut Bergonié, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpitaux civils de Colmar, Colmar
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - IUCT Oncopole, Toulouse
  - lnstitut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No